CLINICAL TRIAL: NCT06364059
Title: A Comparative Analysis of Prognostic Factors for Functional Outcomes in Patients With Acute Subdural Hematoma
Status: Completed | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Military University Hospital, Prague (Other)
Responsible Party: Principal Investigator, Michal Soták, Principal investigator, Charles University, Czech Republic
Other Study IDs: aSDH-TT
Record Dates: First submitted 2024-03-24; First posted 2024-04-15 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Acute Subdural Hematoma; Acquired Brain Injury
Keywords: Acute subdural hematoma; Intracranial hemorrhage; Prognosis; Functional outcome
MeSH Terms: conditions — Hematoma, Subdural, Acute; Brain Injuries; Intracranial Hemorrhages | interventions — Decompressive Craniectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgery Group: Adult patients who underwent surgery due to acute subdural hematoma
  Interventions: Procedure: Decompressive craniectomy with evacuation of subdural hematoma

INTERVENTIONS:
Procedure: Decompressive craniectomy with evacuation of subdural hematoma — Adult patients who underwent decompressive craniectomy with evacuation of subdural hematoma.

SUMMARY:
Acute subdural hematoma (ASDH) is the most common intracranial traumatic lesion that requires surgical intervention. Although there is extensive published research on acute subdural, there remains uncertainty regarding mortality risk and functional outcomes for patients. This study aims to evaluate the effectiveness of contemporary scoring systems in different age groups of ASDH patients to predict functional outcomes.

DETAILED DESCRIPTION:
Acute subdural hematoma (ASDH) is the most common intracranial traumatic lesion that requires surgical intervention. Although there is extensive published research on acute subdural, there remains uncertainty regarding mortality risk and functional outcomes for patients. This study aims to evaluate the effectiveness of contemporary scoring systems in different age groups of ASDH patients to predict functional outcomes. It is our belief that this research will provide valuable insights on the risk of mortality and functional outcomes for ASDH patients. Several clinical and radiologic factors have been identified within the general population that correlate with mortality rates and functional outcomes. There are a number of factors that must be considered in the evaluation of a patient with traumatic brain injury, and a comprehensive assessment is necessary to determine the best course of treatment.

ELIGIBILITY:
Inclusion Criteria:

* surgery due to ASDH
* 12 months of follow-up
* functional outcome measured by the Glasgow Outcome Scale Extended (GOSE).

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who underwent surgery due to acute subdural hematoma in a single institution.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-11-04 (Actual); Study Completion 2025-11-04 (Actual)

PRIMARY OUTCOMES:
Level of consciousness at time of injury | through study completion, an average of 1 year
  The level of consciousness (using the Glasgow Coma Scale, 3-15 points, higher score means a better outcome) at the time of injury is analyzed.
Initial size of subdural hematoma | through study completion, an average of 1 year
  Initial size of subdural hematoma measured in millimetres using CT scan.
Initial midline shift | through study completion, an average of 1 year
  Initial size of midline shift measured in millimetres using CT scan.
Chronic use of anti-clotting medication | once at time of admission
  The number of patients on chronic anticoagulation therapy will be the subject of analysis.
Trauma severity analyzed using Injury Severity Score (ISS). | once at time of admission
  Trauma severity analyzed using Injury Severity Score. The ISS scores ranges from 1 to 75 points (Higher scores correspond to more severe injury and a higher risk of death).
Severity of illness analyzed using Acute Physiology and Chronic Health Evaluation II score (APACHE II) | within 24 hours of admission
  Severity of patient illness will be analyzed using Acute Physiology and Chronic Health Evaluation II score (APACHE II) which ranges from 0 to 71 points. Higher scores correspond to more severe disease and a higher risk of death.
The Glasgow Outcome Scale (GOS) at the time of discharge from the Intensive Care (IC). | through study completion, an average of 1 year
  The Glasgow Outcome Score allowing the objective assessment of the patient´s recovery after trauma brain injury. Allows a prediction of the long-term course of rehabilitation to return to work and everyday life. It uses five categories: 1. Death, 2. Persistent vegetative state, 3. Severe disability, 4. Moderate disability, 5. Low disability.
The Glasgow Outcome Scale Extended (GOSE) evaluation of global disability and recovery after 6 months. | 6 months follow up
  The Glasgow Outcome Scale Extended (GOSE) is an expanded version of the Glasgow Outcome Scale for evaluation of global disability and recovery after traumatic brain injury. It uses eight categories: 1. Death, 2. Vegetative state, 3. Lower severe disability, 4. Upper severe disability, 5. Lower moderate disability, 6. Upper moderate disability - some disability but can potentially return to some form of employment, 7. Lower good recovery - minor physical or mental defect, 8. Upper good recovery - full recovery.
  A GOSE analysis will be performed on a patient who has undergone evacuation of a subdural hematoma 6 months after the trauma.
The Glasgow Outcome Scale Extended (GOSE) evaluation of global disability and recovery after 12 months. | 12 months follow up
  The Glasgow Outcome Scale Extended (GOSE) is an expanded version of the Glasgow Outcome Scale for evaluation of global disability and recovery after traumatic brain injury. It uses eight categories: 1. Death, 2. Vegetative state, 3. Lower severe disability, 4. Upper severe disability, 5. Lower moderate disability, 6. Upper moderate disability - some disability but can potentially return to some form of employment, 7. Lower good recovery - minor physical or mental defect, 8. Upper good recovery - full recovery.
  A GOSE analysis will be performed on a patient who has undergone evacuation of a subdural hematoma 12 months after the trauma.

SECONDARY OUTCOMES:
Number of revisions. | 24 hours
  The number of re-operations that are required within 24 hours of the initial procedure will be analyzed.
Time from injury to surgery. | 24 hours
  The time from the onset of the injury to the evacuation of the subdural hematoma will be analyzed.
Time of operation. | up to 4 hours
  The operative time of the evacuation of the subdural hematoma will be analyzed.
The need for reversal of the effects of anticoagulants. | 24 hours
  The number of cases of need for reversal of the effect of chronic anticoagulant medication will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Tomáš Tyll, M.D., Ph.D., Study Director — Charles University, Czech Republic
Locations (1):
- Military University Hospital Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No